CLINICAL TRIAL: NCT04421963
Title: Roll Over StudY for Patients Who Have Completed a Previous Oncology Study With Olaparib and Are Judged by the Investigator to Clinically Benefit From Continued Treatment
Brief Title: Roll Over StudY for Patients Who Have Completed a Previous Oncology Study With Olaparib
Acronym: ROSY-O
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D0817C00098; 2019-003777-26 (EudraCT Number)
Record Dates: First submitted 2020-05-19; First posted 2020-06-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: HER2-ve metastatic; BRCA mutations; Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Treatment
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — 300 mg olaparib (2×150 mg tablets) twice daily

SUMMARY:
The rationale of the ROSY-O study is to continue to provide study treatment for patients who have participated in a parent study with olaparib and who are continuing to derive clinical benefit from treatment at the end of such studies, as judged by the Investigator.

DETAILED DESCRIPTION:
ROSY-O is an open label, non-randomised, multicentre,international trial for patients who have completed a parent study using olaparib and who are deriving clinical benefit from continued treatment as judged by the Investigator. Patients will be rolled-over from the parent study and will continue the study indefinitely, until they meet one of the treatment discontinuation criteria

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written ICF.
2. Patient is currently deriving clinical benefit, as judged by the Investigator, from continued treatment in an AZ parent study using an AstraZeneca (AZ) compound that has met its endpoints or has otherwise stopped.
3. Patient participating in a prior oncology study with an AZ compound in which they received olaparib and are continuing to receive clinical benefit from treatment; the prior study can be an open-label or blinded study, with unblinding at study close.

Exclusion Criteria:

1. Ongoing, unresolved, Grade 3 or above toxicity requiring interruption of treatment at the time of the termination of the parent study.
2. Currently receiving treatment with any prohibited medication(s).
3. Concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
4. Permanent discontinuation from the parent study due to toxicity or disease progression.
5. Local access to commercially-available drug at no cost to the patient is permitted by local regulation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects with historically diagnosed relapsed high grade serious or high grade endometrioid ovarian cancer; Patients with HER2-ve metastatic breast cancer with germline or somatic BRCA mutations.
Enrollment: 185 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Safety follow up | Baseline up to approximately 10 years
  Serious adverse events and adverse events of special interest reported until 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Locations (89):
- United States (14):
  - Research Site, Boca Raton, Florida
  - Research Site, Towson, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Basking Ridge, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Germantown, Tennessee
  - Research Site, Houston, Texas
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Namur
- Research Site, Rio de Janeiro, Brazil
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (7):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, Changchun, China
- Czechia (4):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Ostrava Poruba
  - Research Site, Prague
- Research Site, Aalborg, Denmark
- Research Site, Kuopio, Finland
- France (4):
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Plérin
  - Research Site, Villejuif
- Research Site, Dresden, Germany
- Research Site, Budapest, Hungary
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (13):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Candiolo
  - Research Site, Catania
  - Research Site, Lecce
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Verona
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Grzepnica
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Research Site, Saint Petersburg, Russia
- Research Site, Ljubljana, Slovenia
- Research Site, Seoul, South Korea
- Spain (10):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Zaragoza
- Research Site, Lund, Sweden
- Research Site, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Şahinbey
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home